CLINICAL TRIAL: NCT02183883
Title: Deciphering Afatinib Response and Resistance With INtratumour Heterogeneity
Acronym: DARWIN1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/14/0131
Record Dates: First submitted 2014-06-27; First posted 2014-07-08 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; Afatinib; Intra-tumour heterogeneity; Clonal dominance; Drug resistance; EGFR; HER2; Phase 2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Afatinib (Experimental): Afatinib, tablet, 40mg, 30mg, 20mg, OD, taken until progression, unacceptable toxicity, intercurrent illness, patient/clinician decision
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — 40mg, 30mg, 20mg, OD, taken until progression, unacceptable toxicity, intercurrent illness, patient/clinician decision.
  EGFR positive mutation patients only: dose escalation to a maximum of 50 mg/day may be considered in patients who tolerate a 40 mg/day dose (i.e. absence of diarrhoea, skin rash, stomatitis, and other adverse reactions with CTCAE Grade > 1) in the first 3 weeks. The dose should not be escalated in any patients with a prior dose reduction. The maximum daily dose for EGFR mutation positive patients is 50 mg.
  Other Names: Giotrif

SUMMARY:
To assess if targeting activating EGFR and HER2 mutations in Non-Small Cell Lung Cancer (NSCLC) is more effective when these mutations are truncal dominant mutations (≥50%), as opposed to non-dominant (≥5 to <50%) or low frequency mutations (<5%).

This trial will be available to patients registered to the TRACERx study (NCT01888601), or non-TRACERx patients who have two archival tissue/DNA samples who are willing to have a biopsy of their relapsed disease.

DETAILED DESCRIPTION:
Increasing evidence suggests that clonal dominance of the drug target should be considered when stratifying therapeutics in solid tumours. It is likely that intratumour heterogeneity and cancer subclonal diversity may contribute to the high failure rate of oncology drugs relative to other medical specialties where drugs are applied to stable somatic genomes rather than unstable genomes found in cancer populations. In addition, increasing evidence in NSCLC and other solid tumours suggests that the selection of resistant subclones during the disease course is responsible for the acquisition of drug resistance and therapeutic failure. Finally, spatial separation of cancer subclones within the same tumour is likely to contribute to the difficulties associated with cancer biomarker validation.

"Actionable mutations" may not be optimally actionable if they are present at one site of disease or within a minority tumour subclone. Such minority subclones are likely to contribute to intratumour heterogeneity and discordant results when interpreting multiple biopsies from the same tumour. Our work in NSCLC, renal cancers and glioblastomas is demonstrating that such subclones, carrying potentially targetable events, may be spatially separated within the same tumour or between primary and metastatic sites. This has been demonstrated in the context of EGFR somatic mutations that may be heterogeneous in up to 25-30% of patients, present at one site of disease but not another. The impact of such actionable driver heterogeneity on treatment response, drug resistance and outcome is currently unclear and is the subject of investigation within this protocol; DARWIN1 will assess the impact of EGFR activating mutation and HER2 mutation heterogeneity on progression free survival outcomes in advanced NSCLC treated with the EGFR tyrosine kinase inhibitor, afatinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing to have a biopsy of relapsed disease. Consent will be obtained through the TRACERx study or with the 'trial entry tissue collection' consent form(non-TRACERx patients). Procurement of the biopsy sample is not necessary at the time of trial registration. However, patients must undergo a biopsy prior to commencement of afatinib.
* Patients must have tumours harbouring a sensitising EGFR mutation or HER2 mutation in at least one biopsy at recurrence, or region of the primary sample.
* Non-TRACERx patients must have at least two archival tissue/DNA samples of their disease available.
* Written informed consent for DARWIN1.
* ECOG performance status 0-3
* No previous exposure to an EGFR TKI (other than afatinib) or HER2 targeted therapy
* Measurable disease by RECIST v1.1. Patients without measurable disease may be eligible following discussion with the CI and UCL CTC but will not count towards the primary PFS endpoint.
* At least 18 years of age.
* Anticipated life expectancy of at least three months.
* Adequate organ function as defined by the following baseline values:

  * Absolute neutrophil count (ANC) ≥1.5x109/L
  * Platelets ≥100x109/L
  * Serum bilirubin ≤1.5 x upper limit of normal (ULN). In patients with known Gilbert's syndrome, total bilirubin ≤3xULN with direct bilirubin ≤1.5xULN
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤3xULN or ≤5x ULN if liver metastases are present
  * Creatinine clearance must be ≥30mL/min
* Women with child-bearing potential, or men who are able to father a child, must be willing to practice highly effective methods of contraception during the trial and for 1 month after the end of treatment.
* Women of childbearing potential must have a negative pregnancy test within 14 days before the first dose of trial medication.

Exclusion Criteria:

* Currently suitable for radical radiotherapy.
* Requirement for intravenous feeding, active peptic ulcer, prior surgical procedures affecting absorption or any medical comorbidity affecting gastrointestinal absorption.
* Patients with current or pre-existing interstitial lung disease.
* Significant or recent acute gastrointestinal abnormalities with diarrhoea as a major symptom e.g. Crohn's disease, malabsorption, or CTCAE v4.03 Grade ≥3 diarrhoea of any etiology at baseline.
* Known hypersensitivity to afatinib or to any of the excipients.
* Patients with rare hereditary conditions of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Women of childbearing potential, or men who are able to father a child, unwilling to use a highly effective method of contraception during the trial.
* Anti-cancer therapy including chemotherapy, immunotherapy, biologic therapy, or major surgery within 14 days prior to start of trial therapy.
* Known human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection. Subjects with evidence of hepatitis B virus clearance may be enrolled.
* History of other malignancy; Exception: (a) Subjects who have been successfully treated and are disease-free for 3 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) CLL in stable remission, or (e) indolent prostate cancer requiring no or only anti-hormonal therapy with histologically confirmed tumor lesions that can be clearly differentiated from lung cancer target and non-target lesions are eligible.
* The following cardiac abnormalities:

  * Corrected QT (QTc) interval ≥480 msecs
  * History of acute coronary syndromes (including unstable angina) within the past 24 weeks
  * Coronary angioplasty, or stenting within the past 24 weeks
  * Class III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * History of known arrhythmias (except sinus arrhythmia) within the past 24 weeks
  * Myocardial infarction within the last 6 months
* Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension etc), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to comply with the requirements of the trial, trial protocol or to provide informed consent.
* Pregnant, lactating or actively breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 60 months
  From date of registration until the date of the last documented progression or date of death from any cause, whichever comes first, assessed up to 60 months.

SECONDARY OUTCOMES:
Overall survival | Up to 60 months
  From date of registration until the date of death from any cause assessed up to 60 months.
Time-to-progression | Up to 60 months
  From date of registration until the date of the last documented progression assessed up to 60 month.
Tumour Response | Up to 60 months
  From date of registration until the date of the last documented response assessed up to 60 months.
Toxicity/Adverse events | Up to 60 months
  Adverse events, including any dose reductions, interruptions and modifications from date of registration up until 60 months.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Forster, Principal Investigator — UCLH
Locations (7):
- United Kingdom (7):
  - Aberdeen Royal Infirmary (NHS Grampian), Aberdeen
  - Barnet and Chase Farm Hospitals (Royal Free London NHS Foundation Trust), Barnet
  - Heart of England NHS Foundation Trust, Birmingham
  - Beatson West of Scotland Cancer Centre (NHS Greater Glasgow & Clyde), Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - Cr Uk & Ucl Ctc, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Danilenko M, Clifford SC, Schwalbe EC. Inter and intra-tumoral heterogeneity as a platform for personalized therapies in medulloblastoma. Pharmacol Ther. 2021 Dec;228:107828. doi: 10.1016/j.pharmthera.2021.107828. Epub 2021 Mar 1. PMID 33662447